CLINICAL TRIAL: NCT05366946
Title: The Prevalence of Chronic Pain in COPD and Its Clinical Implications
Status: Completed | Type: Observational
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Roger Goldstein, Respiratory Physician, West Park Healthcare Centre
Other Study IDs: JREB014
Record Dates: First submitted 2015-10-20; First posted 2022-05-10 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-04

CONDITIONS: COPD
Keywords: Pain
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pain | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- COPD - prevalence: Diagnosed with COPD (based on GOLD criteria and history of > 10 pack years of smoking) and no history of recent musculoskeletal injuries (within last 4 weeks) - prevalence study
  Interventions: Other: Prevalence study
- Healthy controls - prevalence: Not diagnosed with COPD or other respiratory conditions or recent musculoskeletal injuries (within last 4 weeks) - prevalence study
  Interventions: Other: Prevalence study

INTERVENTIONS:
Other: Prevalence study — Prevalence study of chronic pain in COPD vs healthy controls

SUMMARY:
This study explores the prevalence of chronic pain in individuals with COPD compared to healthy controls and examines the clinical implications of pain on symptoms associated with COPD, psychological effect and physical activity.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major public health problem with considerable direct and indirect healthcare costs. COPD is a disease of the older age-group which results in significant disability, high health care costs and is a leading cause of morbidity. This rising disease burden is associated with the systemic effects of this condition, with the clinical presentation of dyspnoea, reduced exercise capacity, fatigue and anxiety all contributing to the reduced health-related quality of life (HRQoL) in people with COPD . In addition to these symptoms, the clinical profile may be further complicated by the presence of pain. Recent studies have found the prevalence of pain ranging from 37 to 72% in COPD, although the duration and frequency of pain experiences across the disease spectrum compared to healthy individuals have not been clearly defined. While chronic pain has been associated with hyperinflation in patients with asthma, the association between pain and lung disease severity, according to spirometry measures and hyperinflation has not been determined in COPD.

According to analysis of body charts, common regions of pain in COPD are the chest, thorax and neck, which are largely similar to healthy populations. However, it is not clear whether the origin of the pain source is musculoskeletal and/or related to postural changes or is due to other sources. Greater exploration of pain within specific spinal regions using well validated tools which focus on musculoskeletal pain will provide further insight into potential causes.

Patients with COPD frequently experience co-morbid conditions which include ischaemic heart disease, diabetes, cancer and musculoskeletal conditions . Although increased pain intensity in COPD appears to be associated with a higher number of co-morbidities, the relationship between co-morbidities and locations of pain, duration, frequency in COPD is not clear. Some concomitant conditions, such as musculoskeletal disorders may influence the prevalence and experience of pain, but this has not been explored in COPD.

In patients with moderate to severe COPD, increased pain severity has been linked to greater interference with activity and a poorer HRQOL. While this provides some insight into the clinical impact of pain, it is equally important to identify the link between pain and other commonly reported symptoms, including dyspnoea. Both pain and dyspnoea are recognised as multidimensional phenomenons, with physiological and psychological consequences and to gain a thorough understanding of each, evaluation of the sensory dimensions (intensity, quality, time course and location) and affective dimensions (unpleasantness and consequent emotional impact) is necessary. Patients with COPD have reported pain with coughing , but the link between the extent of breathlessness, including that experienced during activity and the experience of pain has not been determined. With the shared characteristics and common neural pathways which subserve distress and discomfort in pain and dyspnoea, understanding the relationship between these symptoms may provide further insight into the possible sources of pain in COPD.

To achieve a thorough profile of pain, assessment of the psychosocial impact of pain, including pain catastrophising is recommended. Pain catastrophising is associated with heightened pain experiences, increased levels of disability and depression in non-respiratory conditions and in cystic fibrosis. With anxiety and depression frequently reported in COPD, these clinical symptoms may interact with pain experiences, but the extent to this is unknown.

International guidelines for managing COPD advocate for the role of pulmonary rehabilitation, with compelling evidence of improvement in exercise capacity, reduction in breathlessness and improvement in HRQOL, irrespective of disease severity. As part of this, physical activity is a critical element to disease management. Recently, pain was associated with reduced level of physical activity in those with moderate to severe COPD. However, the relationship between pain locations and the influence upon physical activity is unknown.

Clinical relevance This study aims to impact directly on the important clinical outcomes of HRQOL and disease burden in COPD, markers that are strongly associated with hospitalisation and health care utilisation. Understanding the extent of this comorbidity of pain, its interaction with other symptoms and its broader clinical consequences is the first step in identifying whether modifications to the management of COPD, including the development or institution of therapeutic approaches to minimize pain are necessary. Understanding the psychological consequences of pain in COPD is essential in prioritizing those patients who may require further assessment and treatment of pain.

ELIGIBILITY:
Inclusion Criteria:

* No diagnosis of COPD or other respiratory conditions
* No recent history (within last 4 weeks) of musculoskeletal injury

Exclusion Criteria:

* Diagnosis of other respiratory disease, including COPD
* Recent musculoskeletal injury

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diagnosed with COPD according to GOLD criteria and history of smoking > 10 pack years
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory | Day 1
  Collates information on pain intensity using numerical rating scales, with a higher score denoting greater intensity.
Extended Aberdeen Back Pain Scale (EABPS) | Day 1
  Measure of neck, upper and lower back pain from 35 questions with an overall total score
Self-reported Leeds Assessment of Neuropathic Symptoms and Signs pain scale (S-LANSS) | Day 1
  Consists of 9 items identifying the presence or absence of clinical signs and symptoms with a score of ≥ 12 indicative of neuropathic pain.
Pain Catastrophizing Scale (PCS) | Day 1
  Assesses the presence and extent of catastrophic thoughts or feelings accompanying pain experiences from 13 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Goldstein, MD, Principal Investigator — West Park Healthcare Centre
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada